CLINICAL TRIAL: NCT06360263
Title: OSSEODENSIFICATION BY DENSAH BURS IN COMBINATION WITH ACTIVATED PLASMA ALBUMIN GEL FOR TRANSCRESTAL MAXILLARY SINUS LIFTING WITH SIMULTANEOUS IMPLANT PLACEMENT (CLINICAL TRIAL)
Brief Title: OSSEODENSIFICATION BY DENSAH BURS WITH ACTIVATED PLASMA ALBUMIN GEL FOR SINUS LIFTING WITH SIMULTANEOUS IMPLANT PLACEMENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Esraa Salem Kamal (Other)
Responsible Party: Sponsor-Investigator, Esraa Salem Kamal, Oral and Maxillofacial Surgery MSc Candidate, Alexandria University
Organization: Alexandria University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #1-6/2023
Record Dates: First submitted 2024-04-08; First posted 2024-04-11 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Bone Loss, Alveolar
Keywords: transcrestal sinus lifting
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sinus lifting using densah bur in combination with activated plasma albumin gel (Experimental)
  Interventions: Combination Product: Densah bur in combination with activated plasma albumin gel

INTERVENTIONS:
Combination Product: Densah bur in combination with activated plasma albumin gel — Simultaneous implant placement after transcrestal maxillary sinus lifting using densah burs in combination with activated plasma albumin gel.(APAG). A full mucoperiosteal flap will be elevated, and then reflected with periosteal elevator application of first densah bur (the narrowest) with densifying mood (reverse) counterclockwise, 800-1500 revolutions per minute with copious irrigation until the sinus is reached confirm bur position with a radiograph. Then a wider densah bur (3.0) is used with the same mode and bouncing motion to elevate the sinus floor up to 3 mm in 1mm increments.The sequential densah bur will be used with the same mode and bouncing motion to elevate the the sinus floor 3 mm maximum. After achieving the final planned osteotomy diameter, the osteotomy will be filled with APAG. Then, the desired implant length is inserted.

SUMMARY:
Aim of the current study is to evaluate clinically and radiographically transcrestal sinus lifting with densah burs with the use of activated plasma albumin gel associated with simultaneous implant placement.

ELIGIBILITY:
Inclusion Criteria:

* Patient with missing maxillary premolars and molars.
* Vertical bone height of 3-5 mm.
* Good oral hygiene.
* Non smokers.

Exclusion Criteria:

* Bad oral hygiene.
* Presence of infection or periapical lesions in adjacent teeth.
* Acute maxillary sinusitis.
* Bruxism or clenching.
* Medically compromised patients with a condition that affects the procedure (patients with bone diseases such as osteogenesis imperfecta and polyarthritis and patients on radiotherapy and chemotherapy)

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2023-07-10 (Actual); Primary Completion 2024-07-10 (Actual); Study Completion 2024-07-10 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | up to one week
  This will be assessed using a 10-point Visual Analogue Scale (VAS). (0-1= None, 2-4= Mild, 5-7= Moderate, 8-10= Severe)
Implant stability | up to 6 months
  Resonance frequency analysis is based on determining whether or not an implant is stable enough. The result is presented as an ISQ value of 1-100. The higher the ISQ, the more stable the implant.
Vertical bone height gain | up to 6 months
  To determine the amount of bone height gain, cone beam computed tomography (CBCT) scans will be taken immediately and after 6 months. Amount of bone height gain will be measured linearly in millimeter by determine the difference between residual bone height and bone height above the implant immediately and 6 months postoperatively in anteroposterior and mediolateral dimensions.
Bone density around implant | up to 6 months
  This will be measured from CBCT scans in grayscale using a software. Densitometric analysis will be performed around dental implants on CBCT image using the software supplied with the machine. This analysis gives the actual bone density around the immersed dental implant that proves the process of osseointegration. Higher values indicate better results

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt

REFERENCES:
- [Derived] Kamal ES, Shaaban A, Melek L. Osseodensification by Densah burs in combination with activated plasma albumin gel for transcrestal maxillary sinus lifting with simultaneous implant placement. Oral Maxillofac Surg. 2025 Sep 20;29(1):158. doi: 10.1007/s10006-025-01459-8. PMID 40973834